CLINICAL TRIAL: NCT06914609
Title: Phase 3 Study of the Efficacy and Safety of ION582 in Children and Adults With Angelman Syndrome
Brief Title: REVEAL: A Phase 3 Study of ION582 in Angelman Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ION582-CS2; 2024-519711-33-00 (EU CTIS Number); U1111-1319-2765 (Other: WHO Number)
Record Dates: First submitted 2025-03-22; First posted 2025-04-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Angelman Syndrome
Keywords: ION582; Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 ION582 80 mg (Experimental): Participants (aged 2 to <18 years old) will be administered ION582 80 mg via IT injection Q12W during the double blind and LTE treatment periods.
  Interventions: Drug: ION582
- Cohort 1 Placebo (Placebo Comparator): Participants (aged 2 to <18 years old) will be administered ION582 matching placebo via IT injection Q12W during the double-blind treatment period and then administered ION582 40 mg or 80 mg Q12W during the LTE treatment period.
  Interventions: Drug: Placebo
- Cohort 2 ION582 80 mg (Experimental): Participants (aged 18 to ≤50 years old) will be administered ION582 80 mg via IT injection Q12W during the double blind and LTE treatment periods.
  Interventions: Drug: ION582
- Cohort 2 Placebo (Placebo Comparator): Participants (aged 18 to ≤50 years old) will be administered ION582 matching placebo via IT injection Q12W during the double-blind treatment period and then randomized to ION582 40 mg or 80 mg Q12W during the LTE treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ION582 — ION582 will be administered by IT injection.
  Arms: Cohort 1 ION582 80 mg; Cohort 2 ION582 80 mg
Drug: Placebo — ION582 matching placebo will be administered by IT injection.
  Arms: Cohort 1 Placebo; Cohort 2 Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ION582 in children and adults with Angelman syndrome caused by a deletion or mutation of the UBE3A gene.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled study in people with Angelman syndrome. The study will consist of 4 periods: a screening period of up to 28 days, an approximate 60-week double blind, placebo-controlled treatment period, followed by an approximate 25-month Long-Term Extension (LTE) treatment period, and an approximate 8-month Post-LTE follow-up period. The study will be comprised of 2 cohorts. Cohort 1 will include pediatric participants, aged 2 to less than (<)18 years old and serve as the population for evaluation of primary and secondary outcome measures; Cohort 2 will include adult participants, aged 18 to ≤50 years old. Participants will be randomized 1:1 to 80 mg ION582 or placebo during the double-blind placebo-controlled treatment period. Participants from both cohorts completing the placebo-controlled treatment period will be eligible to transition into the LTE Treatment Period wherein all trial participants will receive ION582. Participant, Caregiver, Investigator and Sponsor will remain blinded to the ION582 dose administered to participants during the LTE.

The study initiated in 2024 with three dosing groups (40 mg ION582, 80 mg ION582, and placebo). Following additional review of data from the ongoing Phase 1/2 trial of ION582 (HALOS), REVEAL was amended in December 2025 to its current form as a two-arm study: 80 mg ION582 and placebo. Following the amendment, participants who were randomized to receive 40 mg ION582 will be transitioned to receive 80 mg ION582.

ELIGIBILITY:
Key Inclusion Criteria:

1. The participants caregiver(s)/ legally authorized representative must have given written informed consent and any authorizations required by local law and be able to comply with all study requirements.
2. Medically stable and can undergo sedation and/or general anesthesia without intubation.
3. Male or female between 2 and lesser than or equal to (≤)50 years of age, depending on specific cohort, at the time of the in-clinic Screening visit.
4. Participant has a clinical diagnosis of Angelman syndrome (AS) with molecular confirmation of either Ubiquitin-protein ligase E3A (UBE3A) deletion or UBE3A mutation.
5. Currently receiving stable doses of concomitant medications typically prescribed for AS, such as anti-epileptic medication, behavioral management medications, sleep medications, gabapentin, cannabidiol, and special diets, supplements, or nutritional support for at least 8 weeks prior to the Baseline visit.
6. Legally authorized representative/caregiver(s) agree(s) not to post any of the participant's personal medical data or information related to the study on any website or social media site (e.g., Facebook, Instagram, X (formerly Twitter), YouTube, TikTok, etc.) from the time of enrollment until they are notified that the study is completed.

Key Exclusion Criteria:

1. Must not have any clinically significant abnormalities in medical history (e.g., major surgery within 3 months of screening), or on physical examination for which treatment with an antisense oligonucleotide (ASO) would be contraindicated or which, in the opinion of the Principal Investigator (PI), could confound the results of this study.
2. Known brain or spinal disease that would interfere with the lumbar puncture (LP) procedure, cerebrospinal fluid (CSF) circulation, or presence of other factors would affect the safety of the LP procedure.
3. Must not have any other conditions, which, in the opinion of the Investigator, would make the participant unsuitable for inclusion or could interfere with the participant participating in or completing the study.
4. Must not have any laboratory abnormalities or any other clinically significant abnormalities that would, as assessed by the Investigator, at screening or Baseline, render a participant unsuitable for inclusion.
5. Previous treatment with an oligonucleotide (including small interfering ribonucleic acid (RNA) [siRNA], ASOs) gene therapy or gene editing. This exclusion criterion does not apply to approved nucleic acid-based vaccines, including mRNA vaccines, which are allowed.
6. Has molecular confirmation of AS due to paternal uniparental disomy, imprinting center defect, or mosaic findings.

Other inclusion/exclusion criteria may apply.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Change in Performance on the Expressive Communication Subdomain Raw Score of the Bayley Scales for Infant and Toddler Development-4 (Bayley-4) Without Caregiver Input in Cohort 1 | Baseline and Week 52
  The Bayley-4 is a performance-based assessment of developmental functioning across communication, cognition, and motor skills. The expressive communication subdomain of communication measures preverbal and verbal communication. The total raw score reflects the sum of all the item scores within the expressive communication subdomain, with higher scores reflecting greater expressive communication ability.

SECONDARY OUTCOMES:
Change in Bayley Scales for Infant and Toddler Development-4 (Bayley-4): Cognition Subdomain Raw Score Without Caregiver Input | Baseline and Week 52
  The Bayley-4 is a performance-based assessment of developmental functioning across communication, cognition, and motor skills. The cognitive subdomain measures learning, memory and concept formation. The total raw score reflects the sum of all the item scores within the expressive communication subdomain, with higher scores reflecting greater cognitive ability.
Change in Symptoms of Angelman Syndrome -Clinician Global Impression of Change (SAS-CGI-C): Overall AS | Baseline and Week 52
  The SAS-CGI-C for Overall AS is a disease-specific clinician-reported outcome assessment measure for Angelman syndrome. The clinicians rate their overall impression of the change of the participant's Angelman syndrome symptoms utilizing a 7-point scale, ranging from "very much improved" (1) to "very much worse" (7).
Change in Vineland Adaptive Behavior Scale-3 (Vineland-3): Receptive Communication Subdomain Raw Score | Baseline and Week 52
  The Vineland-3 assesses adaptive behaviors across 4 domains via a semi-structured interview between a trained clinician and the caregiver of the participant with AS. The receptive communication subdomain of communication measures the participant's ability to attend, understand, and respond appropriately to information from others. The total raw score reflects the sum of all the item scores within the receptive communication subdomain, with higher scores reflecting greater receptive communication ability.
Change in Vineland Adaptive Behavior Scale-3 (Vineland-3): Daily Living Skills, Personal Subdomain Raw Score | Baseline and Week 52
  The Vineland-3 assesses adaptive behaviors across 4 domains via a semi-structured interview between a trained clinician and the caregiver of the participant with AS. The Personal subdomain of the Daily Living Skills domain measures the participant's self-sufficiency in such areas as eating, dressing, washing, hygiene, and health care. The total raw score reflects the sum of all the item scores within the Personal subdomain, with higher scores reflecting greater ability.
Change in Symptoms of Angelman Syndrome - Clinician Global Impression of Change (SAS-CGI-C): Sleep Problems | Baseline and Week 52
  The SAS-CGI-C for Sleep Problems is a disease-specific clinician-reported outcome assessment measure for Angelman syndrome. The clinicians rate their overall impression of the change in the participant's sleep problems utilizing a 7-point scale, ranging from "very much improved" (1) to "very much worse" (7).
Change in Bayley Scales for Infant and Toddler Development-4 (Bayley-4): Fine Motor Subdomain Raw Score Without Caregiver Input | Baseline to Week 52
  The Bayley-4 is a performance-based assessment of developmental functioning across communication, cognition, and motor skills. The Fine Motor subdomain of communication measures motor abilities such as reaching, object manipulation, and grasping. The total raw score reflects the sum of all the item scores within the fine motor subdomain, with higher scores reflecting greater fine motor ability.
Change in Observer-Reported Communication Ability (ORCA): Overall Emerging T Score | Baseline and Week 52
  The ORCA measure assesses, from the caregiver's perspective, the communication ability of individuals with neurodevelopmental disorders, like Angelman syndrome. This questionnaire assesses expressive, receptive, and pragmatic communication. The ORCA measure produces a single score that is an estimate of an individual's overall level of communication ability, with higher T-scores reflecting greater communication ability.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to Week 52
Change in Vital Signs and Clinical Laboratory Results | Baseline and Week 52

CONTACTS AND LOCATIONS:
Locations (24):
- United States (12):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Colorado Children's Hospital Research Institute, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy, Kansas City, Missouri
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill School of Medicine, Carrboro, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Sydney Children's Hospital, Randwick, Australia
- Canada (4):
  - London Health Science Centre - Children's Hospital, London, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - University of Alberta Hospital, Edmonton
  - British Columbia Children's Hospital, Vancouver
- Sheba Medical Center, Ramat Gan, Israel
- Japan (2):
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
- KK Women's and Children's Hospital, Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/